CLINICAL TRIAL: NCT04272697
Title: European Atherosclerosis Society Familial Hypercholesterolaemia Studies Collaboration
Brief Title: EAS Familial Hypercholesterolaemia Studies Collaboration
Acronym: FHSC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 19IC5437
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial hypercholesterolaemia; Primary dyslipidaemia; Cardiovascular disease prevention; LDL cholesterol; Genetic lipids disorders
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heterozygous Familial Hypercholesterolaemia: Adults and children with Heterozygous Familial Hypercholesterolaemia.
- Homozygous Familial Hypercholesterolaemia: Adults and children with Homozygous Familial Hypercholesterolaemia
- Unaffected (non-FH) relatives of FH individuals: Adults and children with unaffected (non-FH) relatives of FH individuals

SUMMARY:
Familial hypercholesterolaemia (FH) is a common genetic disorder resulting in marked elevations in low-density lipoprotein cholesterol (LDL-C). If untreated, lifelong exposure to elevated LDL-C results in a substantially increased risk of (premature) cardiovascular disease as compared to the general population. Although FH adverse cardiovascular outcomes are potentially preventable through early identification of FH individuals and initiation of effective treatment, reports shows that FH is under-diagnosed and under-treated.

Efforts to tackle the global burden of FH have been hindered by a lack of global cohesion, with data held in disparate formats across many sites/countries, resulting in fragmentation and lack of harmonized data from different cohorts. A lack of structure and the availability of limited resources have made it hitherto difficult to integrate these cohorts thus far.

The EAS FHSC is a global initiative of stakeholders involved in the care of people living with FH that seeks to empower the medical and global community to seek changes in their respective countries or organisations to promote early diagnosis and effective treatment of FH. The FHSC Global Registry is a comprehensive, robust database of compiled secondary, unidentifiable, anonymised data on the burden of FH worldwide. These secondary data are sourced from multiple active national/regional/local registries across nearly 60 countries thus far, independent and external to the FHSC, and submitted to the FHSC Registry where data is standardised, pooled, harmonised and integrated into a single global database.

The FHSC Global Registry currently contains over 60,000 cases and remains active and will continue to receive secondary data over the years ahead. This multi-national pooled dataset facilitates clinical observational (non-interventional) studies to address multiple scientific inquires. This hypothesis-free epidemiology research will report on the characteristics of FH worldwide more accurately and inform the development of clinical guidelines and healthcare policy.

DETAILED DESCRIPTION:
Familial hypercholesterolaemia (FH) is a common genetic disorder affecting low-density lipoprotein cholesterol (LDL-C) metabolism, resulting in reduced catabolism of LDL particles and marked elevations in circulating LDL-C. If untreated, lifelong exposure to elevated LDL-C results in the development of atherosclerotic lesions early in life and a substantially increased risk of premature cardiovascular disease as compared to the general population. Early detection and effective treatment of FH can result in a significant improvement in clinical outcomes. Despite these compelling data, FH remains largely underdiagnosed with less than 5% of individuals with FH being identified in most regions around the world. Compounding its burden is the observation that FH is undertreated even among those with an established diagnosis.

The European Atherosclerosis Society (EAS) FH Studies Collaboration (FHSC) is a global initiative that was launched in 2015 to bring together a large-scale consortium of investigators and stakeholders involved in the care of people living with FH. The EAS FHSC ultimately seeks to empower the medical and global community to seek changes in their respective countries or organisations to promote early diagnosis and effective treatment of FH. The Coordinating Centre is based at the Imperial Centre for Cardiovascular Disease Prevention (ICCP), Imperial College London (ICL), UK. Currently investigators from over 65 countries are involved in the EAS FHSC network.

Specifically, the EAS FHSC aims to:

* Establish a worldwide, standardised registry of patients with FH by bringing together regional/national/international cohorts and registries with access to FH patients. This will allow the collaboration to maximise the exploitation of the data to accurately and reliably investigate (i) the burden of both homozygous FH (HoFH) and HeFH, (ii) how FH is detected and managed, (iii) the clinical consequences of current practice on delivery of care and outcomes, (iv) the factors that influence optimal management and LDL-C target attainment in FH.
* Disseminate the information gained from the registry to an international audience including physicians, other healthcare professionals, policy-makers and patients' organizations, to sensitise them to the contemporary burden of FH, encourage open discussion on FH management, promoting a uniform evidence-based standard-of-care, and encourage them to contribute actively to research.
* Consolidate a network of investigators interested in FH through which collaborative research and networking on FH can be conducted on a large-scale.

The FHSC Global Registry is a comprehensive, robust database of compiled secondary, unidentifiable, anonymised data on the burden of FH worldwide. These secondary data were sourced from multiple resources of active multiple cohorts, registries, databases and collections with access to information on individuals with a clinical and/or genetic diagnosis of homozygous or heterozygous FH across nearly 60 countries thus far, independent and external to the FHSC, and submitted to the FHSC Registry by the respective data suppliers where data is pooled, harmonised and integrated into a single global database. The FHSC registry has been conceived with a long term strategy in mind, in order to increase the follow-up of patients, including new individuals diagnosed with FH over time, bringing new cohorts into the registry, and take into account temporal trends and changes in clinical practice.

Quality assurance was addressed by providing the data suppliers with the FHSC protocol, which sets out the criteria of minimal standards for data collection prior to submission to the FHSC Global Registry, ensuring data completeness and accuracy. The incoming data was collated, standardised in accordance with a data dictionary, cleaned and validated by coordinating data queries with the respective data suppliers, and integrated within a secure data warehouse.

The FHSC Global Registry currently contains over 60,000 cases and remains active and will continue to receive secondary data over the years ahead. Standard validated statistical procedures and models for observational studies and weighted meta-analyses are being performed on the secondary data to address multiple scientific inquiries.

Further details, including FHSC protocol, are published open-access at:

FHSC Investigators. Pooling and expanding registries of familial hypercholesterolaemia to assess gaps in care and improve disease management and outcomes: Rationale and design of the global EAS Familial Hypercholesterolaemia Studies Collaboration. Atheroscler Suppl. 2016 Dec;22:1-32. doi: 10.1016/j.atherosclerosissup.2016.10.001.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or genetic diagnosis of heterozygous or homozygous familial hypercholesterolaemia (FH)
* Relatives of index cases without a diagnosis of FH where screening (cascade or other) is carried out.
* The data have been de-identified prior to transferring to the EAS FHSC Global Registry.

Exclusion Criteria:

* Secondary causes of dyslipidaemia (e.g. untreated hypothyroidism, cholestasis, nephrotic syndrome).
* Where data collection does not conform to the local or country wide standards for anonymised data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients clinically and/or genetically diagnosed with familial hypercholesterolaemia (FH).
  Non-affected (non-FH) relatives of FH patients as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2015-03-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Familial Hypercholesterolaemia | Baseline
  Type of FH (Heterozygous FH, Homozygous FH).
  What clinical and/or genetic diagnostic criteria was used to diagnose FH.
  In the case of clinical diagnosis, what criteria system was used (Dutch Lipid Clinics Network, MedPed, Simon-Broome, Japanese [JAS] guidelines criteria, Canadian FH criteria, or other to be specified), what is the likelihood of the diagnosis (possible, probable, definite) and the diagnostic score, and what criteria within the clinical diagnostic system were met (family history of cardiovascular disease [CVD], personal history of premature CVD, physical examination [xanthomas, arcus corneallis], LDL-Cholesterol levels).
  In the case of genetic diagnosis, what gene was affected (LDL receptor, Apolipoprotein B, PCSK9, LDLRAP1, other to be specified).
  Age at diagnosis of FH.
Change in Lipid levels from diagnosis of FH/baseline to follow up | Baseline and follow-up through study completion, average 5 years
  Total cholesterol, LDL-Cholesterol, HDL-Cholesterol, Non-HDL-Cholesterol, Triglycerides, Apolipoprotein A, Apolipoprotien B, Lipoprotein(a)
Characteristics, vascular risk factors and cardiovascular comorbidity associated to FH patients | Baseline
  General and demographic characteristics, including gender, age, ethnicity, and world geographical region.
  Cardiovascular Risk Factors, including hypertension, diabetes (and type I or II), smoking, body mass index, systolic and diastolic blood pressure, and family history of cardiovascular diseases (CVD).
  Cardiovascular Diseases, including coronary artery disease, cerebrovascular disease and peripheral artery disease, and the age at diagnosis (i.e. premature or non-premature CVD).
Change in Management of FH patients over time | Baseline and follow-up through study completion, average 5 years
  Whether patient is on lipid-lowering medication or not. Among those on lipid-lowering medication, what drug, including statins, ezetimibe, PCSK9 inhibitors, other lipid-lowering drugs. In each case, type of drug within each class and dose.
  Proportion of patients who met the guideline-recommended target attainment (LDL-C and non-HDL-C targets, based on the baseline cardiovascular risk) and associated factors.
Risk of adverse outcomes in patients with FH | Through study completion, an average 5 years
  Major Adverse Cardiovascular Events (composite of fatal and non-fatal coronary heart disease, fatal and non-fatal stroke, peripheral vascular disease, and revascularization); Cardiovascular mortality; All-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Ray, MD MPhil, Principal Investigator — Imperial College London
Locations (1):
- School of Public Health, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vallejo-Vaz AJ, Kondapally Seshasai SR, Cole D, Hovingh GK, Kastelein JJ, Mata P, Raal FJ, Santos RD, Soran H, Watts GF, Abifadel M, Aguilar-Salinas CA, Akram A, Alnouri F, Alonso R, Al-Rasadi K, Banach M, Bogsrud MP, Bourbon M, Bruckert E, Car J, Corral P, Descamps O, Dieplinger H, Durst R, Freiberger T, Gaspar IM, Genest J, Harada-Shiba M, Jiang L, Kayikcioglu M, Lam CS, Latkovskis G, Laufs U, Liberopoulos E, Nilsson L, Nordestgaard BG, O'Donoghue JM, Sahebkar A, Schunkert H, Shehab A, Stoll M, Su TC, Susekov A, Widen E, Catapano AL, Ray KK. Familial hypercholesterolaemia: A global call to arms. Atherosclerosis. 2015 Nov;243(1):257-9. doi: 10.1016/j.atherosclerosis.2015.09.021. Epub 2015 Sep 18. No abstract available. PMID 26408930
- [Background] EAS Familial Hypercholesterolaemia Studies Collaboration; Vallejo-Vaz AJ, Akram A, Kondapally Seshasai SR, Cole D, Watts GF, Hovingh GK, Kastelein JJ, Mata P, Raal FJ, Santos RD, Soran H, Freiberger T, Abifadel M, Aguilar-Salinas CA, Alnouri F, Alonso R, Al-Rasadi K, Banach M, Bogsrud MP, Bourbon M, Bruckert E, Car J, Ceska R, Corral P, Descamps O, Dieplinger H, Do CT, Durst R, Ezhov MV, Fras Z, Gaita D, Gaspar IM, Genest J, Harada-Shiba M, Jiang L, Kayikcioglu M, Lam CS, Latkovskis G, Laufs U, Liberopoulos E, Lin J, Lin N, Maher V, Majano N, Marais AD, Marz W, Mirrakhimov E, Miserez AR, Mitchenko O, Nawawi H, Nilsson L, Nordestgaard BG, Paragh G, Petrulioniene Z, Pojskic B, Reiner Z, Sahebkar A, Santos LE, Schunkert H, Shehab A, Slimane MN, Stoll M, Su TC, Susekov A, Tilney M, Tomlinson B, Tselepis AD, Vohnout B, Widen E, Yamashita S, Catapano AL, Ray KK. Pooling and expanding registries of familial hypercholesterolaemia to assess gaps in care and improve disease management and outcomes: Rationale and design of the global EAS Familial Hypercholesterolaemia Studies Collaboration. Atheroscler Suppl. 2016 Dec;22:1-32. doi: 10.1016/j.atherosclerosissup.2016.10.001. Epub 2016 Dec 7. PMID 27939304
- [Background] EAS Familial Hypercholesterolaemia Studies Collaboration; Vallejo-Vaz AJ, De Marco M, Stevens CAT, Akram A, Freiberger T, Hovingh GK, Kastelein JJP, Mata P, Raal FJ, Santos RD, Soran H, Watts GF, Abifadel M, Aguilar-Salinas CA, Al-Khnifsawi M, AlKindi FA, Alnouri F, Alonso R, Al-Rasadi K, Al-Sarraf A, Ashavaid TF, Binder CJ, Bogsrud MP, Bourbon M, Bruckert E, Chlebus K, Corral P, Descamps O, Durst R, Ezhov M, Fras Z, Genest J, Groselj U, Harada-Shiba M, Kayikcioglu M, Lalic K, Lam CSP, Latkovskis G, Laufs U, Liberopoulos E, Lin J, Maher V, Majano N, Marais AD, Marz W, Mirrakhimov E, Miserez AR, Mitchenko O, Nawawi HM, Nordestgaard BG, Paragh G, Petrulioniene Z, Pojskic B, Postadzhiyan A, Reda A, Reiner Z, Sadoh WE, Sahebkar A, Shehab A, Shek AB, Stoll M, Su TC, Subramaniam T, Susekov AV, Symeonides P, Tilney M, Tomlinson B, Truong TH, Tselepis AD, Tybjaerg-Hansen A, Vazquez-Cardenas A, Viigimaa M, Vohnout B, Widen E, Yamashita S, Banach M, Gaita D, Jiang L, Nilsson L, Santos LE, Schunkert H, Tokgozoglu L, Car J, Catapano AL, Ray KK; EAS Familial Hypercholesterolaemia Studies Collaboration (FHSC) Investigators. Overview of the current status of familial hypercholesterolaemia care in over 60 countries - The EAS Familial Hypercholesterolaemia Studies Collaboration (FHSC). Atherosclerosis. 2018 Oct;277:234-255. doi: 10.1016/j.atherosclerosis.2018.08.051. PMID 30270054
- [Derived] European Atherosclerosis Society Familial Hypercholesterolaemia Studies Collaboration. Familial hypercholesterolaemia in children and adolescents from 48 countries: a cross-sectional study. Lancet. 2024 Jan 6;403(10421):55-66. doi: 10.1016/S0140-6736(23)01842-1. Epub 2023 Dec 12. PMID 38101429

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04272697/Prot_SAP_000.pdf